CLINICAL TRIAL: NCT02017509
Title: A Study to Determine the Immunopheotype of Locally Advanced Rectal Adenocarcinoma and Its Correlation With the Efficacy of Neoadjuvant Chemoradiotherapy
Brief Title: Immunoscore in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Providence Health & Services (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: 13-107A
Record Dates: First submitted 2013-12-09; First posted 2013-12-20 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Cancer of the Rectum; Neoplasms, Rectal; Rectal Cancer; Rectal Tumors; Rectal Adenocarcinoma
Keywords: Immunophenotype; Immunoscore; MRI; RNA Later
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients who enroll in the study will all undergo a biopsy as part of their standard of care evaluation. Biopsies samples will be obtained and sent to pathology for paraffin embedded blocks for diagnostic evaluation and for subsequent research. Patients will also have tissue stored in RNA later for subsequent microarray analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal Cancer Patients: Patients with a diagnosis adenocarcinoma of the rectum will provide a tumor sample from their diagnostic biopsy and surgical procedure for research purposes, including RNA gene expression analysis. In addition to a standard MRI, patients will have an Intravoxel Incoherent Motion MRI (IVIM) and a Dynamic Contrast Enhanced MRI (DCE-MRI) for research purposes.
  Interventions: Procedure: Diagnostic Biopsy and Surgical Procedure; Procedure: Intravoxel incoherent motion MRI (IVIM); Procedure: Dynamic Contrast Enhanced MRI (DCE-MRI); Genetic: RNA gene expression analysis

INTERVENTIONS:
Procedure: Diagnostic Biopsy and Surgical Procedure — A tumor sample from the diagnostic biopsy and surgical procedure will be used for research.
Procedure: Intravoxel incoherent motion MRI (IVIM) — At the end of a standard MRI, we will perform IVIM, which is a diffusion-weighted imaging sequence that simultaneously characterizes the microscopic diffusivity of water and the macroscopic transport of water via bulk flow. IVIM may more accurately reflect the properties of the tumor microenvironment including vascular permeability, interstitial fluid pressure, and response to neoadjuvant therapy.
Procedure: Dynamic Contrast Enhanced MRI (DCE-MRI) — Following a standard MRI scan, Dynamic Contrast Enhanced MRI (DCE-MRI) will be done. DCE-MRI is an indicator-dilution experiment in which the delivery and transcapillary transfer of a contrast agent, typically one of a number of gadolinium-based contrast agents (GBCA), is used to assess a number of parameters characterizing tissue physiology. In locally advanced rectal cancer patients, use of DCE-MRI for determining pathologic response has produced equivocal results but more promising data has been published recently in the cervical cancer literature.
Genetic: RNA gene expression analysis — RNA will be collected from biopsy and surgical tissue for gene expression analysis.

SUMMARY:
This is an observational study of tumor samples and MRI imaging in patients with colorectal cancers. A tumor sample, MRI scans, and treatment outcome data will be used for research purposes to see if it is possible to predict patients' response to treatment.

DETAILED DESCRIPTION:
The quality of the immune environment in colorectal cancer biopsy samples correlates with disease-free survival and overall survival more so than current staging conventions. This study will use a scoring system called 'immunoscore' to characterize the immune enviroment. Researchers hypothesize that the immunoscore will correlate with outcomes of colorectal patients treated with neoadjuvant chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a rectal mass suspicious for or known to be an adenocarcinoma of the rectum.
* Age > 18
* Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.

Exclusion Criteria:

* History of other malignancy in the past 2 years except carcinoma in situ of the cervix or bladder, or non-melanomatous skin cancer
* Other medical or psychiatric conditions that in the opinion of the Principal Investigator would preclude safe participation in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of a rectal mass suspicious for or known to be an adenocarcinoma of the rectum.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Correlation of the number of infiltrating leukocytes within a biopsy sample with pathologic response | 16 weeks
  Quantitative immunohistochemical analysis will be performed on parameters of interest on both pre-treatment biopsy specimens as well as post-operative specimens. The pre-treatment sample will be used to establish the immunophenotype score. The primary analysis will evaluate the ability of immunophenotype score to correlate with pathologic response.

CONTACTS AND LOCATIONS:
Overall Officials: Marka Crittenden, MD, PhD, Principal Investigator — Earle A. Chiles Research Institute at Providence Health & Services
Locations (2):
- United States (2):
  - Providence Health & Services, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
This project is being done to contribute pathology samples and patient outcome data to a larger data set intended to validate an algorithm to predict patient outcome based on pathology data obtained at diagnosis. As part of this project, pre-existing samples will be used. There will be new slides made from the samples that will be stained to identify immune response. Pathology analysis and images of the slides will be provided (without patient identifiers) along with de-identified patient outcome data to a central coordinating center.
Supporting Information: Study Protocol
Time Frame: Data made available from study start to study closure (approximately 4 years).
Access Criteria: Only de-identified data will be shared.

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/patients/programs/providence-cancer-center/Pages/default.aspx